CLINICAL TRIAL: NCT02847754
Title: Differentiated Resistance Training of the Paravertebral Muscles in Patients With Unstable Spinal Bone Metastasis Under Concomitant Radiotherapy
Acronym: DISPO-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISPO 2
Record Dates: First submitted 2016-07-12; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Vertebral Bony Metastases
Keywords: bony metastases; physical exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): A patients in arm A carry out daily physical Training consisting of three different isometric exercises under the guidance and supervision of a physiotherapist. Training starts day one (first radiotherapy session), 10 daily units of 30 min each are scheduled during radiotherapy. Patients are expected to continue training until 12 weeks post completion of radiotherapy at home. exercise tailored isometric physical exercise
  Interventions: Other: Isometric resistance training
- B (No Intervention): Patients in arm B (control group) receive 10 daily sessions of 15 min progressive muscle relaxation starting from day one of radiotherapy.

INTERVENTIONS:
Other: Isometric resistance training — Exercises in the "all-fours" position Exercises in the "swimming" Position Exercises in the "forearm support" Position Exercises with elastic "rubber" band
  Arms: A

SUMMARY:
Standard indications for palliative radiation of bony metastases include pain, spinal cord compression, and impending pathologic fractures.

Palliative radiation therapy serves to reduce pain, improve quality of life, and avoid complications. Tailored training of the paravertebral musculature may support Radiation therapy and improve above named factors. DISPO-2 was designed to investigate the impact of tailored physical exercise in patients with unstable vertebral metastases as compared to manual therapy (massage etc.). The trial includes patients with painful unstable bony metastases, patients with spinal cord compression or impending pathological fractures are excluded. The investigations are carried out in a prospective randomized controlled phase-II parallel group design.

DETAILED DESCRIPTION:
Standard indications for palliative radiation of bony metastases include pain, spinal cord compression, and impending pathologic fractures. Palliative radiation therapy serves to reduce pain, improve quality of life, and avoid complications. Tailored training of the paravertebral musculature may support radiation therapy and improve above named factors. DISPO-2 was designed to investigate the impact of tailored physical exercise in patients with unstable vertebral metastases as compared to manual therapy (progressive muscle relaxation). The trial includes patients with painful bony metastases, patients with spinal cord compression or impending pathological fractures are excluded. The investigations are carried out in a prospective randomized controlled phase-II parallel group design.

Patients are randomized to one of the following groups: patients in arm A carry out daily physical training consisting of four different isometric exercises under the guidance and supervision of a physiotherapist. Training starts day one (first radiotherapy session), 10 daily units of 30 min each are scheduled during radiotherapy. Patients are expected to continue training until 12 weeks post completion of radiotherapy at home. Patients in arm B (control group) receive 10 daily sessions of 15 min progressive muscle relaxation starting from day one of radiotherapy. Follow-up of the patients is scheduled at 12 weeks post completion of radiotherapy incl. CT of the spine and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* solitary or multiple vertebral metastases
* thoracic spine
* lumbar spine
* sacrum
* indication for palliative radiation therapy
* age: 18 - 80 years
* Karnofsky index > 70%
* bisphosphonate therapy initiated

Exclusion Criteria:

* bony metastases of cervical spine or pelvis
* impending fracture
* other serious illnesses or medical conditions: therapy-refractory unstable heart disease, congestive heart failure NYHA °III and °IV; coagulopathies
* Significant neurological or psychiatric condition including dementia or seizures or other serious medical condition prohibiting the patient's participation in the trial by judgement of the investigators
* Legal incapacity or limited legal capacity
* Positive serum/ urine beta-HCG/ pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
feasibility of isometric exercise in unstable vertebral bony metastases | 12 weeks post completion of radiotherapy
  completion of all isometric exercises until 12 weeks post RT

SECONDARY OUTCOMES:
progression-free survival (PFS) | 2 years post completion of radiotherapy
  PFS is assessed 2 years post completion of radiotherapy
fracture-free survival (FFS) | 2 years post completion of radiotherapy
  FFS is assessed 2 years post completion of radiotherapy
bone density | 12 weeks post completion radiotherapy
  bone density is assessed 12 weeks post completion of radiotherapy using follow-up CT scan of the spine
pain reduction | Immediately after completion of radiotherapy, 12 and 24 weeks post completion of radiotherapy
  pain is evaluated using the VAS pain scale (0-100 points) at completion and 12/ 24 weeks post completion of radiation
Quality of life | 12 and 24 weeks post completion of therapy
  Quality of life is assessed using the EORTC BM22 questionnaire at 12 and 24 weeks post completion of treatment
Fatigue | 12 and 24 weeks post completion of therapy
  Fatigue is assessed using the EORTC FA13 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Germany, Heidelberg, Germany, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] ABRAMS HL, SPIRO R, GOLDSTEIN N. Metastases in carcinoma; analysis of 1000 autopsied cases. Cancer. 1950 Jan;3(1):74-85. doi: 10.1002/1097-0142(1950)3:13.0.co;2-7. No abstract available. PMID 15405683
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Result] Bubendorf L, Schopfer A, Wagner U, Sauter G, Moch H, Willi N, Gasser TC, Mihatsch MJ. Metastatic patterns of prostate cancer: an autopsy study of 1,589 patients. Hum Pathol. 2000 May;31(5):578-83. doi: 10.1053/hp.2000.6698. PMID 10836297
- [Result] Cheville AL, Girardi J, Clark MM, Rummans TA, Pittelkow T, Brown P, Hanson J, Atherton P, Johnson ME, Sloan JA, Gamble G. Therapeutic exercise during outpatient radiation therapy for advanced cancer: Feasibility and impact on physical well-being. Am J Phys Med Rehabil. 2010 Aug;89(8):611-9. doi: 10.1097/PHM.0b013e3181d3e782. PMID 20531162
- [Result] Harrington KD. Impending pathologic fractures from metastatic malignancy: evaluation and management. Instr Course Lect. 1986;35:357-81. PMID 3819423
- [Result] Murnane A, Geary B, Milne D. The exercise programming preferences and activity levels of cancer patients undergoing radiotherapy treatment. Support Care Cancer. 2012 May;20(5):957-62. doi: 10.1007/s00520-011-1167-z. Epub 2011 Apr 27. PMID 21523349
- [Result] Nikander R, Sievanen H, Ojala K, Oivanen T, Kellokumpu-Lehtinen PL, Saarto T. Effect of a vigorous aerobic regimen on physical performance in breast cancer patients - a randomized controlled pilot trial. Acta Oncol. 2007;46(2):181-6. doi: 10.1080/02841860600833145. PMID 17453366
- [Result] Pilge H, Holzapfel BM, Prodinger PM, Hadjamu M, Gollwitzer H, Rechl H. [Diagnostics and therapy of spinal metastases]. Orthopade. 2011 Feb;40(2):185-93; quiz 194-5. doi: 10.1007/s00132-010-1738-6. German. PMID 21271338
- [Result] Roe JW, Ashforth KM. Prophylactic swallowing exercises for patients receiving radiotherapy for head and neck cancer. Curr Opin Otolaryngol Head Neck Surg. 2011 Jun;19(3):144-9. doi: 10.1097/MOO.0b013e3283457616. PMID 21430531
- [Result] Stevinson C, Fox KR. Feasibility of an exercise rehabilitation programme for cancer patients. Eur J Cancer Care (Engl). 2006 Sep;15(4):386-96. doi: 10.1111/j.1365-2354.2006.00677.x. PMID 16968322
- [Result] Verger E, Salamero M, Conill C. Can Karnofsky performance status be transformed to the Eastern Cooperative Oncology Group scoring scale and vice versa? Eur J Cancer. 1992;28A(8-9):1328-30. doi: 10.1016/0959-8049(92)90510-9. PMID 1515244
- [Result] Zhong H, De Marzo AM, Laughner E, Lim M, Hilton DA, Zagzag D, Buechler P, Isaacs WB, Semenza GL, Simons JW. Overexpression of hypoxia-inducible factor 1alpha in common human cancers and their metastases. Cancer Res. 1999 Nov 15;59(22):5830-5. PMID 10582706
- [Derived] Welte SE, Wiskemann J, Scharhag-Rosenberger F, Forster R, Bostel T, Bruckner T, Schlampp I, Meyerhof E, Sprave T, Nicolay NH, Debus J, Rief H. Differentiated resistance training of the paravertebral muscles in patients with unstable spinal bone metastasis under concomitant radiotherapy: study protocol for a randomized pilot trial. Trials. 2017 Mar 31;18(1):155. doi: 10.1186/s13063-017-1903-x. PMID 28359283